CLINICAL TRIAL: NCT05408416
Title: Comparison of Surgery Outcome Between Preoperative and Intraoperative Intravitreal Injection of Ranibizumab for Vitrectomy in Proliferative Diabetic Retinopathy Patients
Brief Title: Comparison of Surgery Outcome Between Preoperative IVR and Intraoperative IVR in PPV for PDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUPHJinfeng Qu
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: pars plana vitrectomy; ranibizumab; preoperative intravitreal injection; intraoperative intravitreal injection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preoperative group (Active Comparator): PDR patients who received ranibizumab injection (0.5mg/0.05ml) 3-5 days before vitrectomy were assigned to preoperative group
  Interventions: Procedure: preoperative group and intraoperative group
- intraoperative group (Experimental): PDR patients who received ranibizumab injection (0.5mg/0.05ml) at the end of vitrectomy were assigned to intraoperative group
  Interventions: Procedure: preoperative group and intraoperative group

INTERVENTIONS:
Procedure: preoperative group and intraoperative group — ranibizumab injection (0.5mg/0.05ml) 3-5 days before vitrectomy or ranibizumab injection (0.5mg/0.05ml) at the end of vitrectomy

SUMMARY:
Proliferative diabetic retinopathy (PDR) is the most common causes of irreversible blindness in diabetic retinopathy (DR).Intravitreal injection of anti-VEGF drugs is a good adjunct to vitreous surgery for severe PDR. Some studies have confirmed that the application of anti-VEGF drugs before vitrectomy for PDR patients can reduce the difficulty of surgery and improve postoperative best corrected visual acuity (BCVA), but very few researches focused on the injections of anti-VEGF during surgery.Therefore, investigators carry out this clinical trial to compare the effects of preoperative and intraoperative intravitreal injections of ranibizumab (IVR) on vitrectomy outcomes for PDR patients.One group receive ranibizumab injection (0.5mg/0.05ml) 3-5 days before vitrectomy. Another group receive ranibizumab injection (0.5mg/0.05ml) at the end of vitrectomy. Intraoperative and postoperative indices are collected for further comparison.Investigators enroll PDR patients whose baseline characteristics including age, sex, BMI, type of diabetes, HbA1c level, duration of DM, hypertension, previous history of laser photocoagulation, status of lens, indication for surgery, baseline BCVA, IOP, baseline CRT and extent of VAG are comparable.The enrolled eyes are randomly assigned according to the Central Randomization System with a ratio of 1:1 to preoperative IVR group and intraoperative IVR group. Intraoperative including surgery time, intraoperative bleeding, intraocular electrocoagulation use, iatrogenic retinal breaks, relaxing retinotomy and silicone oil tamponade, and postoperative indices including postoperative best-corrected visual acuity (BCVA), central retinal thickness (CRT), postoperative vitreous hemorrhage (VH), neovascular glaucoma (NVG), recurrent retinal detachment, postoperative fibrovascular proliferation progression and reoperationare collected for further comparison.

DETAILED DESCRIPTION:
Proliferative diabetic retinopathy (PDR) is the most common causes of irreversible blindness in diabetic retinopathy (DR).It is characterized by progressive loss of vision, retinal edema, vitreous hemorrhage (VH), retinal neovascularization, fibrovascular proliferation, tractional retinal detachment (TRD) and neovascular glaucoma (NVG).Although pars plana vitrectomy (PPV) is the cornerstone for treatment of advanced PDR, related postoperative complications such as recurrent VH, NVG, and progressive fibrovascular proliferation may still cause serious visual impairment.It is well known that vascular endothelial growth factor (VEGF) is a leading role of the neovascularization, vascular permeability, and diabetic macular edema.Intravitreal injection of anti-VEGF drugs before or during PPV maybe a good adjunct to vitreous surgery for severe PDR. Some studies have confirmed that the application of anti-VEGF drugs before vitrectomy for PDR patients can reduce the difficulty of surgery and improve postoperative best corrected visual acuity (BCVA),but very few researches focused on the injections of anti-VEGF during surgery.Therefore, investigators carried out this study to compare the effects of preoperative and intraoperative intravitreal injections of ranibizumab (IVR) on vitrectomy outcomes for PDR patients.Investigators enroll PDR patients whose baseline characteristics including age, sex, BMI, type of diabetes, HbA1c level, duration of DM, hypertension, previous history of laser photocoagulation, status of lens, indication for surgery, baseline BCVA, IOP, baseline CRT and extent of VAG are comparable.The enrolled eyes are randomly assigned according to the Central Randomization System with a ratio of 1:1 to preoperative IVR group and intraoperative IVR group. Intraoperative and postoperative indices are collected for further comparison. Intraoperative indices including surgery time, intraoperative bleeding, intraocular electrocoagulation use, iatrogenic retinal breaks, relaxing retinotomy and silicone oil tamponade. Investigators compare whether there are statistical differences in the above indicators between the two groups. Meanwhile, postoperative indices are collected during 1week, 1 month, 3 month follow-up, including best-corrected visual acuity (BCVA), central retinal thickness (CRT), postoperative vitreous hemorrhage (VH), neovascular glaucoma (NVG), recurrent retinal detachment, postoperative fibrovascular proliferation progression and reoperation. Investigators compare whether there are statistical differences in the above indicators between the two groups at different visit time.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or more with type 1 or 2 diabetes who were clinically diagnosed with PDR;
* persistent VH for more than 1 month or recurrent VH with or without panretinal photocoagulation (PRP);
* TRD detected by indirect ophthalmoscope or B-scan ultrasonography.

Exclusion Criteria:

* previous vitrectomy or intravitreal injection in the study eyes;
* eyes with any ocular disease that may hinder visual improvement other than PDR, such as optic atrophy or macular hole;
* poor control of diabetes mellitus (DM) with hemoglobin A1c (HbA1c) > 12%;
* history of thromboembolic events (including cerebral vascular infarctions or myocardial infarctions) or coagulation system disorders or receiving anticoagulant or antiplatelet therapy;
* eyes given gas tamponade or additional treatment during follow-up periods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
best-corrected visual acuity (BCVA) | from preoperation to 3 months follow-up
  every visit time
central retinal thickness | from preoperation to 3 months follow-up
  every visit time

SECONDARY OUTCOMES:
surgery time | during surgery
  intraoperative index
intraoperative bleeding | during surgery
  intraoperative index
intraocular electrocoagulation use | during surgery
  intraoperative index
iatrogenic retinal breaks | during surgery
  intraoperative index
relaxing retinotomy | during surgery
  intraoperative index
silicone oil tamponade | during surgery
  intraoperative index
postoperative vitreous hemorrhage | during 3 months follow-up
  postoperative index
neovascular glaucoma | during 3 months follow-up
  postoperative index
recurrent retinal detachment | during 3 months follow-up
  postoperative index
postoperative fibrovascular proliferation progression | during 3 months follow-up
  postoperative index
reoperation | during 3 months follow-up
  postoperative index

CONTACTS AND LOCATIONS:
Overall Officials: Jinfeng Qu, MD, Study Chair — Peking University People's Hospital
Locations (1):
- People's Hospital of Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] He YN, Zhao WH, Bai GY, Fang YH, Zhang J, Yang XG, Ding GG. [Relationship between meat consumption and metabolic syndrome in adults in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2018 Jul 10;39(7):892-897. doi: 10.3760/cma.j.issn.0254-6450.2018.07.006. Chinese. PMID 30060300
- [Background] Tseng VL, Greenberg PB, Scott IU, Anderson KL. Compliance with the American Academy of Ophthalmology Preferred Practice Pattern for Diabetic Retinopathy in a resident ophthalmology clinic. Retina. 2010 May;30(5):787-94. doi: 10.1097/IAE.0b013e3181cd47a2. PMID 20168268
- [Background] Bressler SB, Qin H, Melia M, Bressler NM, Beck RW, Chan CK, Grover S, Miller DG; Diabetic Retinopathy Clinical Research Network. Exploratory analysis of the effect of intravitreal ranibizumab or triamcinolone on worsening of diabetic retinopathy in a randomized clinical trial. JAMA Ophthalmol. 2013 Aug;131(8):1033-40. doi: 10.1001/jamaophthalmol.2013.4154. PMID 23807371
- [Background] Ehrlich R, Harris A, Ciulla TA, Kheradiya N, Winston DM, Wirostko B. Diabetic macular oedema: physical, physiological and molecular factors contribute to this pathological process. Acta Ophthalmol. 2010 May;88(3):279-91. doi: 10.1111/j.1755-3768.2008.01501.x. Epub 2010 Mar 11. PMID 20222885
- [Background] Wang X, Wang G, Wang Y. Intravitreous vascular endothelial growth factor and hypoxia-inducible factor 1a in patients with proliferative diabetic retinopathy. Am J Ophthalmol. 2009 Dec;148(6):883-9. doi: 10.1016/j.ajo.2009.07.007. Epub 2009 Oct 17. PMID 19837381
- [Background] Ferenchak K, Duval R, Cohen JA, MacCumber MW. Intravitreal bevacizumab for postoperative recurrent vitreous hemorrhage after vitrectomy for proliferative diabetic retinopathy. Retina. 2014 Jun;34(6):1177-81. doi: 10.1097/IAE.0000000000000058. PMID 24457977
- [Background] Comyn O, Wickham L, Charteris DG, Sullivan PM, Ezra E, Gregor Z, Aylward GW, da Cruz L, Fabinyi D, Peto T, Restori M, Xing W, Bunce C, Hykin PG, Bainbridge JW. Ranibizumab pretreatment in diabetic vitrectomy: a pilot randomised controlled trial (the RaDiVit study). Eye (Lond). 2017 Sep;31(9):1253-1258. doi: 10.1038/eye.2017.75. Epub 2017 May 12. PMID 28498374
- [Background] Simunovic MP, Maberley DA. ANTI-VASCULAR ENDOTHELIAL GROWTH FACTOR THERAPY FOR PROLIFERATIVE DIABETIC RETINOPATHY: A Systematic Review and Meta-Analysis. Retina. 2015 Oct;35(10):1931-42. doi: 10.1097/IAE.0000000000000723. PMID 26398553
- [Background] di Lauro R, De Ruggiero P, di Lauro R, di Lauro MT, Romano MR. Intravitreal bevacizumab for surgical treatment of severe proliferative diabetic retinopathy. Graefes Arch Clin Exp Ophthalmol. 2010 Jun;248(6):785-91. doi: 10.1007/s00417-010-1303-3. Epub 2010 Feb 5. PMID 20135139
- [Background] Ren X, Bu S, Zhang X, Jiang Y, Tan L, Zhang H, Li X. Safety and efficacy of intravitreal conbercept injection after vitrectomy for the treatment of proliferative diabetic retinopathy. Eye (Lond). 2019 Jul;33(7):1177-1183. doi: 10.1038/s41433-019-0396-0. Epub 2019 Mar 14. PMID 30872770
- [Derived] Li S, Tang J, Han X, Wang Z, Zhang L, Zhao M, Qu J. Prospective Comparison of Surgery Outcome Between Preoperative and Intraoperative Intravitreal Injection of Ranibizumab for Vitrectomy in Proliferative Diabetic Retinopathy Patients. Ophthalmol Ther. 2022 Oct;11(5):1833-1845. doi: 10.1007/s40123-022-00550-7. Epub 2022 Jul 29. PMID 35904708